CLINICAL TRIAL: NCT06417944
Title: The Effect of Three-dimensional Exercise (Schroth Exercise) on Diaphragm Thickness in Adolescent Idiopathic Scoliosis Patients
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 326
Record Dates: First submitted 2024-04-28; First posted 2024-05-16 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-04

CONDITIONS: Spine Deformity; Scoliosis; Scoliosis Idiopathic; Scoliosis; Adolescence; Diaphragm Issues
Keywords: Adolescent Idiopathic Scoliosis; Diaphragm Thickness; Three-dimensional Exercise (Schroth Exercise); Ultrasonographic Measurement
MeSH Terms: conditions — Scoliosis | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Schroth group (Group 1): Patients aged 10-18 years who are diagnosed with scoliosis and given 10 sessions of schroth exercises, either outpatient or inpatient.
  Scoliosis study forms consisting of clinical and radiological measurements of patients aged 10-18 years who applied to the outpatient clinic with spine deformity will be filled in in detail.
  Interventions: Diagnostic Test: Scoliosis study form; Diagnostic Test: Scoliosis X-ray (orthorontgenogram); Diagnostic Test: Pulmonary function test; Diagnostic Test: Ultrasonographic Measurement; Procedure: Three-dimensional Exercise (BSPTS Schroth Exercise)
- Control group (Group 2): Patients aged 10-18 years who are diagnosed with scoliosis and given home exercise Scoliosis study forms consisting of clinical and radiological measurements of patients aged 10-18 years who applied to the outpatient clinic with spine deformity will be filled in in detail.
  Interventions: Diagnostic Test: Scoliosis study form; Diagnostic Test: Scoliosis X-ray (orthorontgenogram); Diagnostic Test: Pulmonary function test; Diagnostic Test: Ultrasonographic Measurement; Procedure: Home Exercise

INTERVENTIONS:
Diagnostic Test: Scoliosis study form — Scoliosis study form consisting of clinical and radiological measurements of patients aged 10-18 years who applied to the outpatient clinic with spine deformity will be filled in detail.
Diagnostic Test: Scoliosis X-ray (orthorontgenogram) — Patients whose Adam's forward bending test and clinical evaluation results are compatible with scoliosis, scoliosis graphy are requested. (Adams test (forward bending test) (+) was measured by Bunnell scoliometer (scoliosis assessment tool) and ATR (angle of trunk rotation angle) values were 5 degrees in those with BMI (Body Mass Index) above 85%. If it is below 85% and above 7 degrees, patients who meet the inclusion criteria will be included in the study by filling out an informed consent form and a scoliosis film will be requested.).Coronal, sagittal balance; coronal and sagittal Cobb angles will be measured from posterior-anterior (PA) and lateral scoliosis radiographs.
Diagnostic Test: Pulmonary function test — Pulmonary function tests (PFTs) are noninvasive tests that show how well the lungs are working. The tests measure lung volume, capacity, rates of flow, and gas exchange. This information can help your healthcare provider diagnose and decide the treatment of certain lung disorders. We will use handheld spirometry device for measurement. Three measurements will be made. In these three measurements; FEV1(Forced Expiratory Volume In One Second)(L), FEV1 (%predicted), FVC (Forced Vital Capacity) (L), FVC (%predicted), FEV1/FVC (%) and FEV1/FVC (%predicted) will be evaluated. The arithmetic average of the results of these three measurements will be taken.
  Other Names: Spirometry Function Test
Diagnostic Test: Ultrasonographic Measurement — Diaphragm thickness will be measured in the supine position with a 6-14 Mhz lineer, conventional ultrasound probe (Mindray DC-8, Shenzen Mindray Bio-Medical Electronics CO. LTD.,P.R. China) at the end of inspiration and expiration from the intercostal space on the anterior axillary line. The measurements will be evaluated by making three measurements from the right 8-9. intercostal space where the diaphragm is best visualized. End-expiratory (Forced residual capacity-FRC) (centimeter- cm), end-inspiratory (Total Lung Capacity) (centimeter-cm) and thickening rate (%) (thickness TLC / thickness FRC) will be evaluated three times and the arithmetic average of these three measurements will be taken.
Procedure: Three-dimensional Exercise (BSPTS Schroth Exercise) — It only provides outpatient treatment, but it has different practices, intensive or regular, depending on local and external patients. For local patients, it is applied once a week, accompanied by a therapist, and the treatment duration is determined according to the patient's condition. In patients coming from outside; It can be continued as 2 hours a day for 10 days, then as additional treatment for 1-2 weeks for 3-6 months depending on the patient's condition. I In regular treatment; 30 sessions of 90 minutes group treatment, the first 8 sessions are carried out under the supervision of a therapist for a shorter period of time.
  We will give 10 sessions of BSPTS Schroth exercises, either outpatient or inpatient. After 10 sessions of the Schroth exercise program, the home program will continue two months after outpatient/inpatient schroth exercise(Home program: 5 days/week, 45-60 minutes for all patients).
  Other Names: Physiotherapy Scoliosis Specific Exercises -PSSE (SOSORT Guidelines)
  Groups: Schroth group (Group 1)
Procedure: Home Exercise — In the home exercise program; daily living activities, neutral pelvis exercises, coronal balance exercises, rotational angular breathing exercises and axial elongation exercises were taught by the physiotherapist in one session. A total of 10-week home exercise program was planned, with exercises to be performed twice a week for the first two weeks, once every 15 days for 1 month (twice in one month), and then once a month.
  Groups: Control group (Group 2)

SUMMARY:
Spinal deformity is common in childhood and adolescence, and can often present as scoliosis or increased thoracic kyphosis deformity with various etiologies.The diaphragm is the main respiratory muscle, and diaphragm contraction is associated with respiratory functions.Any spinal deformity, especially one that affects the thoracic spine, can affect lung function.In the planned thesis study, investigators will measure the diaphragm thickness in adolescent idiopathic scoliosis patients with scoliosis deformities affecting the thoracic region, whether there is any relationship between the impact in the thoracic region and the diaphragm thickness, and the three-dimensional exercise (Schroth exercise-Barcelona Schroth therapy) applied in investigators' clinic for scoliosis, before and after the treatment of the diaphragm. Investigators aimed to show whether there is any change in thickness.

DETAILED DESCRIPTION:
Spinal deformity is common in childhood and adolescence, and can often present as scoliosis or increased thoracic kyphosis deformity with various etiologies.

Any spinal deformity, especially one that affects the thoracic spine, can affect lung function. If left untreated, the curves may distort over time as skeletal growth accelerates. In some patients, this can lead to restrictive or obstructive lung disease and, rarely, death as a result of cor pulmonale.

The alignment of the skeletal system in the chest and its harmony with the compliance of the chest wall are related to respiratory function; Thoracic kyphosis and the resulting changes in the rib cage lead to a decrease in lung capacity. The diaphragm is the main respiratory muscle, and diaphragm contraction is associated with respiratory functions. In recent years, ultrasonography (USG) has gained increasing utility for visualizing the diaphragm and assessing its function, with several advantages.

In the planned thesis study, investigators will measure the diaphragm thickness in adolescent idiopathic scoliosis patients with scoliosis deformities affecting the thoracic region, whether there is any relationship between the impact in the thoracic region and the diaphragm thickness, and the three-dimensional exercise (Schroth exercise-Barcelona Schroth therapy) applied in investigators' clinic for scoliosis, before and after the treatment of the diaphragm. Investigators aimed to show whether there is any change in thickness.

ELIGIBILITY:
Inclusion Criteria:

* Having scoliosis affecting the thoracic region according to BSPTS (type 3C, type 4C and its subtypes)
* Being between the ages of 10-18
* Being able to perform a respiratory function test
* Having the mental capacity to answer surveys

Exclusion Criteria:

* Congenital spinal, costal and diaphragmatic anomalies
* Neuromuscular disease
* Respiratory system diseases that affect lung functions
* Patients who cannot cooperate with spirometry.
* Having surgery to the chest wall or spine

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Demographic information of all individuals included in the study will be collected. According to the Barcelona Scoliosis Physical Therapy School (BSPTS) Classification by Rigo and Weiss, the diaphragm thickness in patients diagnosed with scoliosis (type 3C and 4C) with thoracic curvature and in the control group was measured in the supine position with a 7-13 Mhz linear conventional ultrasound probe (brand) on the anterior axillary line. It will be measured at the end of inspiration and expiration from the intercostal space. Three measurements will be made on the right side and the arithmetic average will be evaluated. Follow-up measurement will be made by the same person, with the same device and with the same method in the 3rd month after the treatment.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Scoliosis study form | Within 2 week of applying to the scoliosis outpatient clinic
  Scoliosis study form consisting of clinical and radiological measurements of patients aged 10-18 years who applied to the outpatient clinic with spine deformity will be filled in detail.
Pulmonary function test | Within 2 weeks after applying to the scoliosis clinic (pre-exercise) and 3 months after exercise
  We will use handheld spirometry device for measurement. Three measurements will be made. In these three measurements; FEV1(Forced Expiratory Volume In One Second) (Liter-L), FEV1 (%predicted), FVC (Forced Vital Capacity) (Liter-L), FVC (%predicted), FEV1/FVC (%) and FEV1/FVC (%predicted) will be evaluated. The arithmetic average of the results of these three measurements will be taken.
Ultrasonographic Diaphragm Thickness Measurement | Within 2 weeks after applying to the scoliosis clinic(pre-exercise) and 3 months after exercise
  Diaphragm thickness (millimeter-mm) will be measured in the supine position with a 6-14 Mhz lineer, conventional ultrasound probe (Mindray DC-8, Shenzen Mindray Bio-Medical Electronics CO. LTD.,P.R. China) at the end of inspiration and expiration from the intercostal space on the anterior axillary line. The measurements will be evaluated by making three measurements from the right 8-9. intercostal space where the diaphragm is best visualized. Diaphragm thickness of End-expiratory (Forced residual capacity-FRC) (millimeter-mm), diaphragm thickness of end-inspiratory (Total Lung Capacity) (millimeter-mm) and thickening rate (%) (thickness TLC / thickness FRC) will be evaluated three times and the arithmetic average of these three measurements will be taken.

SECONDARY OUTCOMES:
The Pediatric Quality of Life Inventory | Within 2 weeks after applying to the scoliosis clinic(pre-exercise) and 3 months after exercise
  The Pediatric Quality of Life Inventory (PedsQL) is a 23-item generic health status instrument with parent and child forms that assesses five domains of health (physical functioning, emotional functioning, psychosocial functioning, social functioning, and school functioning) in children and adolescents ages 2 to 18. Each item of the instrument is scored on a 5-point scale from 0- 4 for ages 8-18, (0 = never a problem, 1 = almost never a problem, 2 = sometimes a problem, 3 = often a problem, 4 = almost always a problem) ad 3-point scale for young child self reporting (ages 5- 7) as following (0 = not at all a problem, 2 = sometimes a problem, 4 = a lot of a problem) the large score means worst symptoms , scores are linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0) in which high score means better condition
Scoliosis Research Society Score | Within 2 weeks after applying to the scoliosis clinic(pre-exercise) and 3 months after exercise
  The SRS-22r is a validated questionnaire intended to assess outcomes in patients with idiopathic scoliosis after spinal surgery. The first version, developed by the Scoliosis Research Society in 1999, had 24 items, and this was reduced to 22 items (accompanied by a name change) in the course of 3 major updates.The SRS-22 contains 22 questions covering 5 domains: function/activity 5 items; pain 5 items; self-perceived image 5 items; mental health 5 items; and satisfaction with treatment 2 items. Each item is scored from 1 (worst) to 5 (best). Each domain has a total sum score ranging from 5 to 25, except for satisfaction, which ranges from 2 to 10. The sum of the first 4 domains gives a maximum subtotal of 100, and when the satisfaction domain is included, the maximum total is 110

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Metin Terzibasioglu, MD,Chief Assistant, Study Chair — Maltepe District, Askeri Firin Street, Inistanbul buildins F1 Block Flat: 82 Zeytinburnu /ISTANBUL; Ebru Yilmaz Yalcinkaya, MD,Professor, Study Director — Gaziosmanpaşa Training and Research Hospital Physical Rehabilitation Department
Locations (1):
- Omer Faruk Alp, Istanbul, Gaziosmanpasa, Turkey (Türkiye)

REFERENCES:
- [Background] Jagger F, Tsirikos AI, Blacklock S, Urquhart DS. Adaptation to reduced lung function in children and young people with spinal deformity. J Clin Orthop Trauma. 2020 Mar-Apr;11(2):191-195. doi: 10.1016/j.jcot.2019.12.013. Epub 2020 Jan 3. PMID 32099278
- [Result] Karaali E, Ciloglu O, Gorgulu FF, Ekiz T. Ultrasonographic measurement of diaphragm thickness in patients with severe thoracic scoliosis. J Ultrasound. 2021 Mar;24(1):75-79. doi: 10.1007/s40477-020-00536-w. Epub 2021 Feb 7. PMID 33550575